CLINICAL TRIAL: NCT06257641
Title: Impact of the Mediterranean Diet on Patients with Psoriasis: a Randomized Clinical Trial
Brief Title: Impact of the Mediterranean Diet on Patients with Psoriasis
Acronym: MEDIPSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Javier Pérez Bootello, Principal Investigator, Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEDIPSO
Record Dates: First submitted 2024-01-21; First posted 2024-02-14 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis; Psoriasis Vulgaris; Hyperlipidemias; Depression; Anxiety; Metabolic Syndrome; Obesity
Keywords: Psoriasis; Mediterranean diet; Dietary intervention; Psoriasis vulgaris; Metabolic syndrome
MeSH Terms: conditions — Psoriasis; Hyperlipidemias; Depression; Anxiety Disorders; Metabolic Syndrome; Obesity

STUDY DESIGN:
Intervention Model Description: Experimental, randomised, controlled, open-label, single-blind (outcome assessor) study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-intensity Mediterranean diet (Experimental): Patients assigned to the intervention group will undergo dietary education for the adoption of the Mediterranean diet, with monthly monitoring - mostly online - by nutritionists with experience in the field. Patients will be given 500 ml of extra virgin olive oil per week and informative material about the Mediterranean diet, as well as recipes and weekly menus.
  Interventions: Other: High-intensity Mediterranean diet intervention
- Standard of care (No Intervention): Patients assigned to the control group will be provided with standard recommendations for a low-fat diet with no monitoring by nutritionists.

INTERVENTIONS:
Other: High-intensity Mediterranean diet intervention — Dietary education for the adoption of the Mediterranean diet, with monthly monitoring - mostly online - by nutritionists with experience in the field. Patients will be given 500 ml of extra virgin olive oil per week and informative material about the Mediterranean diet, as well as recipes and weekly menus.
  Arms: High-intensity Mediterranean diet

SUMMARY:
The goal of this clinical trial is to determine the effect of a high-intensity Mediterranean diet intervention over 16 weeks in a group of patients with mild to moderate psoriasis in terms of skin improvement as measured by PASI. In addition, the aim of this study will be to gather the necessary information for a larger and more extended clinical trial in the future.

Participants will be provided with dietary education for the implementation of the Mediterranean diet, supported by a monthly follow-up by nutritionists with experience in the field. Researchers will compare the effect of the Mediterranean diet on these patients to a control group provided with standard recommendations for a low-fat diet with no monitoring by nutritionists.

DETAILED DESCRIPTION:
MEDIPSO is an experimental, randomised, controlled, open-label, single-blinded (evaluator) study. It is a clinical trial in which patients with mild to moderate psoriasis with stable topical treatment are randomly assigned to either the control group or the intervention group. Patients assigned to the intervention group will undergo dietary education for the adoption of the Mediterranean diet, with monthly monitoring - mostly online - by nutritionists with experience in the field. In both groups, blood tests with metabolic parameters will be obtained before and after the study period, and data of anthropometric characteristics and quality of life will be assessed. The effect of the intervention on skin involvement, metabolic parameters and inflammatory cytokines will be assessed, and the emotional and quality of life impact will also be investigated. In addition, a methodological analysis will be carried out in order to improve the design for a larger scale clinical trial in the future.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis clinically diagnosed by a dermatologist.
* Predominantly psoriasis vulgaris.
* Psoriasis Area and Severity Index (PASI) ≥2 and ≤ 10 at the time of recruitment.
* Stable weight (< 5% weight loss or gain) in the last 3 months.
* Treated exclusively with topical treatment for psoriasis at enrolment and throughout the study.
* Able to give informed consent.
* Willing and able to follow the study procedure.
* Willing and able to attend all scheduled visits during the study period.
* Willing and able to provide blood samples as indicated in the procedure.
* Willing to implement pregnancy prevention measures throughout the study period.

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus.
* Good adherence to the Mediterranean diet at the time of screening (er-MEDAS ≥8).
* Language barrier (patients not fluent in Spanish or English).
* Conditions that make telephone communication difficult (e.g. severe hearing loss).
* History of cardiac disease(s).
* Comorbidities that may compromise the implementation of the intervention (e.g. cancer, digestive diseases...) or limit survival to less than 6 months.
* History or current eating disorder (anorexia, bulimia, etc.; screening will be carried out using the Diagnostic and Statistical Manual of Mental Disorders, fifth edition, if indicated).
* Malnourished patients (screening using the Malnutrition Universal Screening Tool -MUST-, if indicated).
* Presenting gout.
* Pregnant, planning pregnancy or breastfeeding.
* Use of diuretics at the time of sampling.
* BMI greater than 40 kg/m2.
* Difficulty or inconvenience in changing dietary habits and following the Mediterranean diet (allergies, food intolerances, special diets).
* Participation in a clinical trial with drugs or dietary intervention in the year prior to inclusion in this study.
* Patients who during the recruitment period are expected to have poor collaboration, lack of commitment or real difficulties in following the development of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Psoriasis Area and Severity Index (PASI) at week 16 | Baseline and week 16
  The Psoriasis Area Severity Index (PASI) is the most widely used scale for assessing the severity of psoriasis and for therapeutic decision making. It ranges from 0 (no lesions) to 72 (worst possible lesions throughout all body surface).

SECONDARY OUTCOMES:
Change from baseline in weight at week 16 | Baseline and week 16
  Weight in kilograms will be assessed by a physician at baseline and week 16
Change from baseline in body mass index (BMI) at week 16 | Baseline and week 16
  BMI in kg/m^2 will be assessed by a physician at baseline and week 16
Change from baseline in abdominal circumference at week 16 | Baseline and week 16
  Abdominal circumference in centimetres will be assessed by a physician at baseline and week 16
Change from baseline in serum inflammatory interleukins at week 16 | Baseline and week 16
  Change in levels of Granulocyte-macrophage colony-stimulating factor (GM-CSF), interferon gamma (IFNγ), interleukin 1β (IL-1β), IL 2, IL 4, IL 5, IL 6, IL 9, IL 10, IL 12 (p70), IL 13, IL 15, IL 17A/CTLA8, IL-17E/ IL-25, IL 17F, IL 21, IL 22, IL 23, IL 27, IL 28A/IFNλ2, IL 31, IL 33/NF HEV (mature), MIP-3α/CCL20, tumoral necrosis factor alpha (TNFα) and TNFβ/Lymphotoxin-α (LTA), all of them measured in pg/ml will also be assessed.
Change from baseline in serum lipids at week 16 | Baseline and week 16
  Change in levels of serum cholesterol, low-density lipoproteins (LDL), high-density lipoproteins (HDL), lipoprotein A, apolipoprotein A1, apolipoprotein B1 measured in mg/dl will also be assessed.
Change from baseline in fasting serum insulin levels at week 16 | Baseline and week 16
  Change in levels of fasting serum insulin levels measured in µUl/ml will also be assessed.
Change from baseline in glycated haemoglobin at week 16 | Baseline and week 16
  Change in levels of glycated haemoglobin measured in percentage (%) will also be assessed.
Change from baseline in C reactive protein at week 16 | Baseline and week 16
  Change in levels of C reactive protein measured in mg/L will also be assessed.
Change from baseline in adherence to mediterranean diet at week 16 | Baseline and week 16
  Change in adherence to mediterranean diet will be assessed by the validated questionnaire energy-restricted Mediterranean Diet Adherence Screener (er-MEDAS), which ranges from 0 to 17 (higher score means better adherence to Mediterranean diet)
Change from baseline in quality of life at week 16 | Baseline and week 16
  Change in quality of life will be assessed by the validated questionnaire Dermatology Life Quality Index (DLQI), which ranges from 0 to 30 (higher score means worse quality of life)
Change from baseline in quality of sleep at week 16 | Baseline and week 16
  Change in quality of sleep will be assessed by the validated questionnaire Insomnia Severity Index (ISI), which ranges from 0 to 28 (higher score means more severe insomnia)
Change from baseline in emotional state at week 16 | Baseline and week 16
  Change in emotional state will be assessed by the validated questionnaire Hospital Anxiety and Depression Scale (HADS). It consists of two sub-scales for Anxiety and Depression, both of which range from 0 to 21 (higher score means more severe anxiety/depression symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Pérez Bootello, Principal Investigator — Hospital Universitario Ramón y Cajal. Instituto Ramón y Cajal de Investigación Sanitaria
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be published as soon as possible, and the overall results will be published when the study finishes and all data is collected.
Supporting Information: Study Protocol, CSR
Time Frame: The study protocol will be published as soon as possible, and the overall results will be published when the study finishes and all data is collected.
Access Criteria: All the information will be open access

REFERENCES:
- [Background] Di Meglio P, Villanova F, Nestle FO. Psoriasis. Cold Spring Harb Perspect Med. 2014 Aug 1;4(8):a015354. doi: 10.1101/cshperspect.a015354. PMID 25085957
- [Background] Kocic H, Damiani G, Stamenkovic B, Tirant M, Jovic A, Tiodorovic D, Peris K. Dietary compounds as potential modulators of microRNA expression in psoriasis. Ther Adv Chronic Dis. 2019 Aug 7;10:2040622319864805. doi: 10.1177/2040622319864805. eCollection 2019. PMID 31431821
- [Background] Castaldo G, Rastrelli L, Galdo G, Molettieri P, Rotondi Aufiero F, Cereda E. Aggressive weight-loss program with a ketogenic induction phase for the treatment of chronic plaque psoriasis: A proof-of-concept, single-arm, open-label clinical trial. Nutrition. 2020 Jun;74:110757. doi: 10.1016/j.nut.2020.110757. Epub 2020 Feb 5. PMID 32222582
- [Background] Tuttolomondo A, Simonetta I, Daidone M, Mogavero A, Ortello A, Pinto A. Metabolic and Vascular Effect of the Mediterranean Diet. Int J Mol Sci. 2019 Sep 23;20(19):4716. doi: 10.3390/ijms20194716. PMID 31547615
- [Background] Phan C, Touvier M, Kesse-Guyot E, Adjibade M, Hercberg S, Wolkenstein P, Chosidow O, Ezzedine K, Sbidian E. Association Between Mediterranean Anti-inflammatory Dietary Profile and Severity of Psoriasis: Results From the NutriNet-Sante Cohort. JAMA Dermatol. 2018 Sep 1;154(9):1017-1024. doi: 10.1001/jamadermatol.2018.2127. PMID 30046840
- [Background] Caso F, Navarini L, Carubbi F, Picchianti-Diamanti A, Chimenti MS, Tasso M, Currado D, Ruscitti P, Ciccozzi M, Annarumma A, Lagana B, Perricone R, Afeltra A, Giacomelli R, Scarpa R, Costa L. Mediterranean diet and Psoriatic Arthritis activity: a multicenter cross-sectional study. Rheumatol Int. 2020 Jun;40(6):951-958. doi: 10.1007/s00296-019-04458-7. Epub 2019 Oct 11. PMID 31605152
- [Background] Martinez-Gonzalez MA, Salas-Salvado J, Estruch R, Corella D, Fito M, Ros E; PREDIMED INVESTIGATORS. Benefits of the Mediterranean Diet: Insights From the PREDIMED Study. Prog Cardiovasc Dis. 2015 Jul-Aug;58(1):50-60. doi: 10.1016/j.pcad.2015.04.003. Epub 2015 May 1. PMID 25940230
- [Background] Goni L, de la O V, Barrio-Lopez MT, Ramos P, Tercedor L, Ibanez-Criado JL, Castellanos E, Ibanez Criado A, Macias Ruiz R, Garcia-Bolao I, Almendral J, Martinez-Gonzalez MA, Ruiz-Canela M. A Remote Nutritional Intervention to Change the Dietary Habits of Patients Undergoing Ablation of Atrial Fibrillation: Randomized Controlled Trial. J Med Internet Res. 2020 Dec 7;22(12):e21436. doi: 10.2196/21436. PMID 33284131
- [Background] Berna-Rico E, Fernandez-Nieto D, Gonzalez-Cantero A. RF - Role of the Mediterranean Diet in the Treatment of Psoriasis. Actas Dermosifiliogr. 2023 Feb;114(2):152-155. doi: 10.1016/j.ad.2021.11.011. Epub 2022 Aug 10. No abstract available. English, Spanish. PMID 35963333
- [Background] Schroder H, Fito M, Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Lamuela-Raventos R, Ros E, Salaverria I, Fiol M, Lapetra J, Vinyoles E, Gomez-Gracia E, Lahoz C, Serra-Majem L, Pinto X, Ruiz-Gutierrez V, Covas MI. A short screener is valid for assessing Mediterranean diet adherence among older Spanish men and women. J Nutr. 2011 Jun;141(6):1140-5. doi: 10.3945/jn.110.135566. Epub 2011 Apr 20. PMID 21508208
- [Background] Schroder H, Zomeno MD, Martinez-Gonzalez MA, Salas-Salvado J, Corella D, Vioque J, Romaguera D, Martinez JA, Tinahones FJ, Miranda JL, Estruch R, Bueno-Cavanillas A, Alonso Gomez AM, Tur JA, Warnberg J, Serra-Majem L, Martin V, Vazquez C, Lapetra J, Pinto X, Vidal J, Daimiel L, Gaforio JJ, Matia-Martin P, Ros E, Lassale C, Ruiz-Canela M, Babio N, Sorli JV, Garcia-Arellano A, Diaz-Lopez A, Fito M, Castaner O; PREDIMED-Plus investigators. Validity of the energy-restricted Mediterranean Diet Adherence Screener. Clin Nutr. 2021 Aug;40(8):4971-4979. doi: 10.1016/j.clnu.2021.06.030. Epub 2021 Jul 6. PMID 34364236
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Fito M, Gea A, Hernan MA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts. N Engl J Med. 2018 Jun 21;378(25):e34. doi: 10.1056/NEJMoa1800389. Epub 2018 Jun 13. PMID 29897866
- [Derived] Perez-Bootello J, Berna-Rico E, Abbad-Jaime de Aragon C, Goni L, Vazquez-Ruiz Z, Neria F, Cova-Martin R, Naharro-Rodriguez J, Ballester-Martinez A, Pindado-Ortega C, Monge D, Blauvelt A, Jaen P, Mehta N, Gelfand JM, Martinez-Gonzalez MA, Gonzalez-Cantero A. Mediterranean Diet and Patients With Psoriasis: The MEDIPSO Randomized Clinical Trial. JAMA Dermatol. 2025 Dec 1;161(12):1215-1223. doi: 10.1001/jamadermatol.2025.3410. PMID 40991259
- [Derived] Perez-Bootello J, Berna-Rico E, Abbad-Jaime de Aragon C, Cova-Martin R, Goni L, Ballester-Martinez A, Jaen-Olasolo P, Mehta N, Gelfand JM, Martinez-Gonzalez MA, Gonzalez-Cantero A. Impact of the Mediterranean Diet on Patients With Psoriasis: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jan 29;14:e64277. doi: 10.2196/64277. PMID 39879606